CLINICAL TRIAL: NCT02870309
Title: Phase I/II Multicenter, Open-label Trial to Evaluate the Safety and Pharmacokinetics of Alpha-1 MP in Patients With Alpha1-Antitrypsin Deficiency
Brief Title: Safety and Pharmacokinetics of Alpha-1 MP (Alpha1-proteinase Inhibitor (Human), Modified Process) in Participants With Alpha1-Antitrypsin Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Grifols Japan K.K. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI1401; JapicCTI-163160 (Other: JapicCTI)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — Mp alpha1 receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Alpha-1 MP (Experimental): Participants received 8 IV infusions of 60 mg/kg Alpha-1 MP administered weekly at an infusion rate not exceeding 0.08 mL/kg/min over approximately 15 minutes, up to Week 8.
  Interventions: Biological: Alpha-1 MP

INTERVENTIONS:
Biological: Alpha-1 MP — Alpha-1 MP is a stable, sterile, lyophilized preparation of human alpha1-PI, also known as α1-antitrypsin
  Other Names: Prolastin-C

SUMMARY:
This study is a multicenter, open-label trial to evaluate the safety and pharmacokinetics of weekly intravenous infusions of 60 mg/kg of Alpha-1 MP (alpha1-proteinase inhibitor (human), modified process) for 8 weeks.

DETAILED DESCRIPTION:
This study is a multicenter, open-label trial to evaluate the safety and pharmacokinetics of weekly intravenous (IV) infusions of 60 mg/kg of the investigational drug in participants with alpha1-antitrypsin deficiency (AATD). The trial will be conducted at approximately 5 medical institutions in Japan, aiming to enroll a minimum of 3 adult participants or more. The trial will consist of a screening period scheduled within 3 weeks before trial entry, an open-label treatment period for 8 weeks, and a pharmacokinetic (PK) evaluation period for 1 week. At the Week 9 visit when the PK evaluation period is completed, participant will be asked whether they would like to participate in an extension trial (GTI1401-OLE). For participants not intending to participate in the extension trial, the date of follow-up/study completion visit (30 days [4 weeks] after the last dose of the investigational drug) will be arranged. Participants will participate in this trial for approximately 14 weeks from the start of the screening period through the completion of the trial.

At the screening visit (scheduled within 3 weeks before trial entry), after providing informed consent (agreement based on adequate explanation and understanding of the treatment plan), participants will be evaluated for eligibility for participation during the screening period. Participants considered eligible will enter the 8-week treatment period to receive a total of 8 weekly IV infusions of 60 mg/kg of Alpha-1 MP. The initial IV infusion will be given at the Week 1 (baseline) visit. During the treatment period, participants will receive weekly IV infusions of Alpha-1 MP at the Weeks 1 (baseline), 2, 3, 4, 5, 6, 7, and 8 visits. After the last IV infusion of Alpha-1 MP at the Week 8 visit, participants will enter the 1-week PK evaluation period. During this PK evaluation period, participants will visit the study center to undergo blood sampling for PK evaluation at the PK1 visit (the next day of the Week 8 visit), the PK2 visit (2 days after the Week 8 visit), the PK5 visit (5 days after the Week 8 visit), and at the Week 9 visit. At 30 days after the last dose (Week 8), participants will visit the study center for follow-up/study completion (Week 12). All participants will undergo blood sampling for the measurement of alpha1-PI trough concentrations at the Weeks 1 (baseline), 7, and 8 visits (blood samples will be collected before dosing) as well as at the Week 9 visit.

Blood samples for the evaluation of PK parameters will be collected from Week 8 to Week 9. The blood sample collected before the infusion of Alpha-1 MP at the Week 8 visit and the blood sample for PK evaluation collected at the Week 9 visit (7 days after the infusion at the Week 8 visit) will be also used for the measurement of alpha1-PI trough concentrations for Weeks 8 and 9.

At the Week 9 visit, participants will be asked whether they would like to participate in the extension trial (GTI1401-OLE). Participants intending to participate in the extension trial will be able to continue the treatment with IV infusions of 60 mg/kg of Alpha-1 MP for at least another year (participants will be further asked whether they would like to continue the treatment at yearly intervals) for the purpose of evaluation of the safety of long-term Alpha-1 MP treatment. Participants not intending to enter the extension trial will visit the study center for follow-up/study completion at 30 days (4 weeks) after the last dose of Alpha-1 MP (Week 12).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥20 years at the time of providing informed consent.
* Participants with clinically apparent pulmonary emphysema diagnosed by Computed Tomography (CT) scan.
* AATD participants with documented serum alpha1-PI levels of <50 mg/dL (i.e., 11 µM) as measured by nephelometry. In participants with no previously documented serum alpha1-PI levels, their serum alpha1-PI levels measured by nephelometry during the screening period must be <50 mg/dL.
* Participants whose percentage of forced expired volume in 1 second/forced vital capacity forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) after inhalation of a bronchodilator is <70% during the screening period [equivalent to the criterion for the diagnosis of chronic obstructive pulmonary disease (COPD)].
* Participants who are willing to and able to provide signed written informed consent.

Exclusion Criteria:

* Participants with moderately or severely deteriorated lung function in the 4 weeks before the Week 1 (baseline) visit.
* Participants whose percentage of forced expired volume in 1 second/forced vital capacity (%FEV1 after inhalation of a bronchodilator is <30% during the screening period.
* Participants who have undergone lung transplantation or liver transplantation.
* Participants who have undergone any lung surgery (excluding lung biopsy) in the past 2 years.
* Participants with increased liver enzymes aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase (AST, ALT, and ALP) ≥2.5 times the upper limit of normal.
* Participants with severe complications including but not limited to congestive heart failure and liver cirrhosis.
* Participants who have developed any malignant tumor (including malignant melanoma; however, other forms of skin cancer are excluded) in the past 5 years.
* Pregnant women, breastfeeding women, or women of childbearing potential who do not intend to use effective contraceptive methods (use of oral, injection, or implant hormonal contraceptives; placement of an intrauterine device (IUD) or intrauterine contraceptive system; concomitant use of spermatocidal foam, gel, film, cream, suppository and condoms or cervical caps; male sterilization; or abstinence) throughout the trial period or male participants who have a partner who is of childbearing potential and is unwilling to use effective contraceptive methods throughout the trial period.
* Participants with a past history of hepatitis A virus, hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HAV, HBV, HCV, or HIV) infection, or participants currently presenting with clinical signs or symptoms suggestive of such infection.
* Participants with a smoking history in the past 6 months, or participants tested positive for urinary cotinine levels at the screening visit.
* Participants participating in another clinical trial within 4 weeks before the Week 1 (baseline) visit.
* Participants with a history of anaphylactic or severe systemic reactions to any plasma derived alpha1-PI product or other blood products.
* Participants who have continuously received any systemic steroid therapy at a prednisone-equivalent dose >5 mg/day within 4 weeks before the Week 1 (baseline) visit (Note: inhaled steroids are not regarded as systemic steroids).
* Participants who have used any systemic or aerosolized antibiotic drug for the treatment of COPD exacerbation within 4 weeks before the Week 1(baseline) visit.
* Participants with a previous or current diagnosis of selective, severe Immunoglobulin A (IgA) deficiency.
* Participants who are mentally challenged and cannot independently give consent.
* Participants who have difficulty in adhering to the protocol or its procedures in the opinion of the investigator.
* Participants who have medical conditions that may confound the results of this clinical trial or may endanger other participants during the participation in this clinical trial in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Hokkaido University Hospital, Sapporo
  - Juntendo University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seyama K, Nukiwa T, Sato T, Suzuki M, Konno S, Takahashi K, Nishimura M, Steinmann K, Sorrells S, Chen J, Hayashi KI. Safety and pharmacokinetics of Alpha-1 MP (Prolastin(R)-C) in Japanese patients with alpha1-antitrypsin (AAT) deficiency. Respir Investig. 2019 Jan;57(1):89-96. doi: 10.1016/j.resinv.2018.09.006. Epub 2018 Nov 8. PMID 30416054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 2 medical institutions in Japan from 29 July 2016 to 15 March 2017.
Period: Overall Study
Arm/Group | Alpha-1 MP
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether considered related to the medicinal product. TEAEs were defined as any AE occurring after or on the first Alpha-1 MP infusion until the final visit of study.
Time Frame: Up to Week 12
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 3

2. Primary Outcome: Number of Participants With Adverse Drug Reaction (ADRs)
Description: ADRs were defined as adverse events (AEs) which were in the investigator's opinion of causal relationship to the study treatment. AE was defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product.
Time Frame: Up to Week 12
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 1

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Week 12
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

4. Primary Outcome: Number of Discontinuations Due to Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether considered related to the medicinal product. TEAEs were defined as any AE occurring after or on the first Alpha-1 MP infusion until the final visit of study. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Week 12
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

5. Primary Outcome: Number of Participants With Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: COPD exacerbation was defined as an increase in respiratory symptoms (dyspnea, increased cough, and/or production of sputum) over baseline that usually requires medical intervention.
Time Frame: Up to Week 12
Population: Safety population included all the participants who received any amount of Alpha-1 MP.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Trough Level of Total alpha1-PI for Weekly IV Infusions of 60 mg/kg Alpha-1 MP
Time Frame: Baseline (Week 1), Weeks 7, 8 (prior to the start of infusions of Alpha-1 MP) and Week 9 (168 hours post infusion)
Population: Pharmacokinetic (PK) population included all the participants who received Alpha-1 MP dose and had sufficient samples to calculate the PK parameters. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: milligram/decilitre
Arm/Group | Alpha-1 MP
Number analyzed (Participants) | 4
milligram/decilitre
  Week 1 | 11.450 (3.5162)
  Week 7: number analyzed (Participants) | 3
  Week 7 | 55.567 (7.2231)
  Week 8 | 55.425 (7.2325)
  Week 9 | 56.900 (12.9378)

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the end of study (Up to Week 12).
Arm/Group | Alpha-1 MP
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha-1 MP (N=4)
Fatigue (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT02870309/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT02870309/SAP_001.pdf